CLINICAL TRIAL: NCT06512701
Title: Study on the Correlation Between Fat Soluble Vitamins and Non-alcoholic Fatty Liver Disease
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Liu Zhong, Clinical Professor, First Affiliated Hospital of Zhejiang University
Other Study IDs: 20240727
Record Dates: First submitted 2024-07-10; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Fat Soluble Vitamin Deficiencies and Disorders
Keywords: cross-sectional study; correlation; dose-response relationship
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:  — This study is an observational study without any intervention measures.

SUMMARY:
Excessive or insufficient levels of vitamins in the body can affect health. With the prevalence of obesity and MetS, NAFLD has become the leading cause of chronic liver disease and abnormal liver biochemical indicators in health examinations in China. The current research results on serum vitamin A, D, and E levels in NAFLD patients are controversial. Therefore, this study mainly explores the correlation between serum FSV levels and NAFLD, providing reference for nutrition and clinical management of NAFLD patients.

DETAILED DESCRIPTION:
This is a single center cross-sectional study. In this study, 4000 eligible patients will be recruited and demographic information and clinical data of all study subjects will be collected. According to the results of abdominal ultrasound, the patients were divided into NAFLD group and non NAFLD group. The levels of fat soluble vitamins in the two groups were compared to explore the correlation between different concentrations of fat soluble vitamin levels and the risk of NAFLD.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, both male and female;
2. Voluntarily participate in this study and sign an informed consent form;
3. Diagnosed NAFLD through abdominal ultrasound;

Exclusion Criteria:

1. Acute and chronic infections, severe cardiovascular and cerebrovascular diseases, respiratory system diseases, urinary system diseases, rheumatic diseases, tumors, and pituitary dysfunction; Or have hepatitis B, hepatitis C virus, or acquired immunodeficiency syndrome;
2. Surgery was performed within 6 months, and blood donation, transfusion, or significant blood loss occurred within 4 months;
3. Have taken vitamin supplements within 2 weeks;
4. Women are in pregnancy, lactation, or within one year after childbirth;
5. Alcohol abuse (alcohol intake ≥ 140 g/week for males and ≥ 70 g/week for females)
6. The serum creatinine (SCr) exceeds twice the following abnormal values, with the standard of abnormal values being: male (20-59 years old)>97 μ mol/L, male (60-79 years old)>111 μ mol/L; Female (20-59 years old)>73 μ mol/L, female (60-79 years old)>81 μ mol/L.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 and above who underwent physical examinations at the Health Management Center of the First Affiliated Hospital of Zhejiang University School of Medicine from July 2024 to June 2026.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-10 (Estimated)

PRIMARY OUTCOMES:
non-alcoholic fatty liver disease prevanlence | Day 1
serum vitamin A | Day 1
serum vitamin D | Day 1
serum vitamin E | Day 1
serum vitamin k | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Liu, MD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No